CLINICAL TRIAL: NCT00152451
Title: An Open-label, Exploratory, Multicenter, Dose-escalation Study Examining the Efficacy, Safety and Tolerability of Ucb 44212 Used at Doses of 10 mg, 20 mg, 40 mg and 80 mg b.i.d. (Total Daily Dose of 20 to 160 mg) in Adult Subjects (18-65 Years) With Refractory Epilepsy Suffering From Partial Onset Seizures (Whether or Not Secondarily Generalized) and Treated With 1, 2 or 3 Approved Antiepileptic Drugs
Brief Title: Study With Seletracetam (Ucb 44212) in Adult Subjects (18 to 65 Years) With Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB S.A. - Pharma Sector (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01191
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-09

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy; Partial onset seizures; Seletracetam
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Seletracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Seletracetam (Experimental): Escalating doses twice daily were to be administered.
  Interventions: Drug: Seletracetam (ucb 44212)

INTERVENTIONS:
Drug: Seletracetam (ucb 44212) — * Pharmaceutical form: oral capsules
  * Concentration: 10 and 50 mg
  * Route of administration: oral administration

SUMMARY:
This trial will evaluate the efficacy and safety of ucb 44212 as add on therapy in subjects with focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Males/Females from 18 to 65 years of age (minimum body weight of 40 kg)
* Subjects with a confirmed diagnosis of epilepsy suffering from partial onset seizures whether or not secondarily generalized
* Subjects who have been treated for epilepsy for >=6 months and are currently uncontrolled while being treated with 1-3 concomitant Antiepileptic Drug (AEDs)
* Female subjects without childbearing potential; Female subjects with childbearing potential are eligible if they use a medically accepted non-hormonal contraceptive method

Exclusion Criteria:

* Seizures occurring in clusters.
* Status epilepticus within 6 months of Visit 1
* History of non-epileptic seizures
* Subjects on vigabatrin
* Subjects on felbamate, unless treatment has been continuous for >2 years
* Ongoing psychiatric disease other than mild controlled disorders.
* Subjects with clinically significant organ dysfunction
* Known allergic reaction or intolerance to pyrrolidine derivatives and/or excipients
* Pregnant or lactating women
* Subjects currently taking levetiracetam (LEV)
* Use of benzodiazepines (for any indication) taken at a higher frequency than an average of once a week, unless counted as one of the concomitant Antiepileptic Drug (AEDs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-05-19 (Actual); Primary Completion 2006-05-03 (Actual); Study Completion 2006-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (7):
- United States (7):
  - N01191 108, Little Rock, Arkansas
  - N01191 105, San Francisco, California
  - N01191 102, Stanford, California
  - N01191 107, Columbus, Ohio
  - N01191 104, Philadelphia, Pennsylvania
  - N01191 101, Nashville, Tennessee
  - N01191 103, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in May 2005 and concluded in May 2006.
Pre-assignment Details: Participant Flow refers to the Intention-To-Treat Set. The study consisted of a 4-week Baseline Period, a 11-week Treatment Period (Up-/Down-Titration) and a 2-week Post-Treatment Period. Patients were up-titrated every two weeks until the maximum tolerated dose was reached. They were maintained at this dose until the end of the 8-week Up-Titration Period and continue that dose until the Down-Titration Visit scheduled for that dose level. Patients were to be down-titrated over a 3-week Period.
Groups:
- Seletracetam: Escalating doses of 10, 20, 40 and 80 mg b.i.d. (twice daily) (total daily doses of 20 - 160 mg) were to be administered orally as capsules.
Period: Overall Study
Arm/Group | Seletracetam
Started | 31
Completed | 27
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-To-Treat (ITT) Set which consisted of all subjects who took at least one dose of trial medication.
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.41 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Seizure Frequency Per Week of Partial Onset Seizures (Type I) During the Up-titration Period
Description: Calculated as (7-day seizure frequency during the up-titration period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)), divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in partial onset seizure frequency from Baseline.
  The duration of the Up-Titration Period was 8 weeks (Visit 3/Week 5 to Visit 7/Week 12).
Time Frame: During the Up-titration Period (Week 5 to Week 12), compared to Baseline Period (Week 1 to Week 4)
Population: The intention-to-treat (ITT) set included 31 subjects, who took at least one dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
percentage of change | -30.88 [-50.00 to -15.38]

2. Secondary Outcome: Percentage Change From Baseline in Seizure Frequency Per Week of Partial Onset Seizures (Type I) by Visit Over the Treatment Period (Up-titration + Down-titration)
Description: Calculated as (7-day seizure frequency during the Treatment Period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)), divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in partial onset seizure frequency from Baseline.
  The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15). Visit x includes the period from the beginning of Visit x-1 up to but not including Visit x.
Time Frame: During the Treatment Period (Week 5 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication. Only subjects with valid data for partial (Type I) seizure frequency per week at the respective visit are included in the analysis. Number of participants analyzed is given separately per visit.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
percentage of change
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 30
  Visit 4 (Week 5 and 6) | -40.06 [-68.75 to 1.73]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 27
  Visit 5 (Week 7 and 8) | -37.50 [-51.79 to -0.75]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 27
  Visit 6 (Week 9 and 10) | -27.68 [-53.12 to -14.29]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 30
  Visit 7 (Week 11 and 12) | -39.88 [-70.83 to -24.37]
  Visit 8 (Week 13): number analyzed (Participants) | 27
  Visit 8 (Week 13) | -39.33 [-56.76 to -1.69]
  Visit 9 (Week 14): number analyzed (Participants) | 27
  Visit 9 (Week 14) | -41.67 [-61.19 to 25.00]
  Visit 10 (Week 15): number analyzed (Participants) | 27
  Visit 10 (Week 15) | -33.33 [-83.07 to 58.65]

3. Secondary Outcome: Percentage Change From Baseline in Seizure Frequency Per Week for Partial Onset Seizures (Type I) Overall in the Down-titration Period
Description: Calculated as (7-day seizure frequency during the down-titration period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)), divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in partial onset seizure frequency from Baseline.
  The duration of the Down-Titration Period was 3 weeks (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: During the Down-Titration Period (Week 13 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication. Only subjects with valid data for partial (Type I) seizure frequency per week in the down-titration period are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 27
percentage of change | -36.36 [-64.29 to 21.81]

4. Secondary Outcome: Percentage Change From Baseline in Seizure Frequency Per Week for All Seizure Types (Types I+II+III) by Visit Over the Treatment Period (Up-titration + Down-titration)
Description: Calculated as (7-day seizure frequency during the Treatment Period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)), divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in seizure frequency from Baseline.
  The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15). Visit x includes the period from the beginning of Visit x-1 up to but not including Visit x.
Time Frame: During the Treatment Period (Week 5 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication. Only subjects with valid data for all types (Type I+II+III) seizure frequency per week at the respective visit are included in the analysis. Number of participants analyzed is given separately per visit.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
percentage of change
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 30
  Visit 4 (Week 5 and 6) | -40.06 [-68.75 to 3.29]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 27
  Visit 5 (Week 7 and 8) | -37.50 [-51.79 to -0.75]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 27
  Visit 6 (Week 9 and 10) | -27.68 [-53.12 to -14.29]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 30
  Visit 7 (Week 11 and 12) | -39.88 [-70.83 to -24.37]
  Visit 8 (Week 13): number analyzed (Participants) | 27
  Visit 8 (Week 13) | -39.33 [-56.76 to -1.69]
  Visit 9 (Week 14): number analyzed (Participants) | 27
  Visit 9 (Week 14) | -41.67 [-61.19 to 25.00]
  Visit 10 (Week 15): number analyzed (Participants) | 27
  Visit 10 (Week 15) | -33.33 [-83.07 to 58.65]

5. Secondary Outcome: Percentage Change From Baseline in Seizure Frequency Per Week for All Seizure Types (Types I+II+III) Overall in the Up-titration Period
Description: Calculated as (7-day seizure frequency during the up-titration period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)), divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in seizure frequency from Baseline.
  The duration of the Up-Titration Period was 8 weeks (Visit 3/Week 5 to Visit 7/Week 12).
Time Frame: During the Up-Titration Period (Week 5 to Week 12), compared to Baseline Period (Week 1 to Week 4)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
percentage of change | -30.88 [-50.00 to -15.38]

6. Secondary Outcome: Percentage Change From Baseline in Seizure Frequency Per Week for All Seizure Types (Types I+II+III) Overall in the Down-titration Period
Description: Calculated as (7-day seizure frequency during the down-titration period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)), divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in seizure frequency from Baseline.
  The duration of the Down-Titration Period was 3 weeks (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: During the Down-Titration Period (Week 13 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication. Only subjects with valid data for all types (Type I+II+III) seizure frequency per week in the down-titration period are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 27
percentage of change | -36.36 [-64.29 to 21.81]

7. Secondary Outcome: Seizure Frequency Per Week for Partial Onset Seizures (Type I) by Visit Over the Treatment Period
Description: Calculated as 7-day partial onset seizure (type I) frequency; The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15). Visit x includes the period from the beginning of Visit x-1 up to but not including Visit x.
Time Frame: During the Treatment Period (Week 5 to Week 15)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 30
  Visit 4 (Week 5 and 6) | 2.50 [1.00 to 10.50]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 27
  Visit 5 (Week 7 and 8) | 3.73 [1.00 to 13.00]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 27
  Visit 6 (Week 9 and 10) | 2.55 [1.50 to 13.50]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 30
  Visit 7 (Week 11 and 12) | 2.50 [0.88 to 8.62]
  Visit 8 (Week 13): number analyzed (Participants) | 27
  Visit 8 (Week 13) | 3.00 [1.00 to 13.00]
  Visit 9 (Week 14): number analyzed (Participants) | 27
  Visit 9 (Week 14) | 4.00 [2.00 to 13.22]
  Visit 10 (Week 15): number analyzed (Participants) | 27
  Visit 10 (Week 15) | 4.38 [1.75 to 14.00]

8. Secondary Outcome: Seizure Frequency Per Week for Partial Onset Seizure (Type I) Overall in the Treatment Period
Description: Calculated as 7-day partial onset seizure (type I) frequency. The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: During the Treatment Period (Week 5 to Week 15)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week | 2.74 [1.71 to 11.76]

9. Secondary Outcome: Seizure Frequency Per Week for Partial Onset Seizure (Type I) Overall in the Up-titration Period
Description: Calculated as 7-day partial onset seizure (type I) frequency. The duration of the Up-Titration Period was 8 weeks (Visit 3/Week 5 to Visit 7/Week 12).
Time Frame: During the Up-Titration Period (Week 5 to Week 12)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week | 2.25 [1.63 to 9.82]

10. Secondary Outcome: Seizure Frequency Per Week for Partial Onset Seizure (Type I) Overall in the Down-titration Period
Description: Calculated as 7-day partial onset seizure (type I) frequency. The duration of the Down-Titration Period was 3 weeks (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: During the Down-Titration Period (Week 13 to Week 15)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 27
seizures per week | 3.50 [1.75 to 13.70]

11. Secondary Outcome: Seizure Frequency Per Week for All Seizure Types (Type I+II+III) by Visit Over the Treatment Period
Description: Calculated as 7-day seizure frequency for all seizure types (type I+II+III). The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15). Visit x includes the period from the beginning of Visit x-1 up to but not including Visit x.
Time Frame: During the Treatment Period (Week 5 to Week 15)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 30
  Visit 4 (Week 5 and 6) | 2.50 [1.00 to 10.50]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 27
  Visit 5 (Week 7 and 8) | 3.73 [1.00 to 13.00]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 27
  Visit 6 (Week 9 and 10) | 2.55 [1.50 to 13.50]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 30
  Visit 7 (Week 11 and 12) | 2.50 [0.88 to 8.62]
  Visit 8 (Week 13): number analyzed (Participants) | 27
  Visit 8 (Week 13) | 3.00 [1.00 to 13.00]
  Visit 9 (Week 14): number analyzed (Participants) | 27
  Visit 9 (Week 14) | 4.00 [2.00 to 13.22]
  Visit 10 (Week 15): number analyzed (Participants) | 27
  Visit 10 (Week 15) | 4.38 [1.75 to 14.00]

12. Secondary Outcome: Seizure Frequency Per Week for All Seizure Types (Type I+II+III) Overall in the Treatment Period
Description: Calculated as 7-day seizure frequency for all seizure types (type I+II+III). The Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: During the Treatment Period (Week 5 to Week 15)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week | 2.74 [1.71 to 11.76]

13. Secondary Outcome: Seizure Frequency Per Week for All Seizure Types (Type I+II+III) Overall in the Up-titration Period
Description: Calculated as 7-day seizure frequency for all seizure types (type I+II+III). The duration of the Up-Titration Period was 8 weeks (Visit 3/Week 5 to Visit 7/Week 12).
Time Frame: During the Up-Titration Period (Week 5 to Week 12)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication.
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week | 2.25 [1.63 to 9.82]

14. Secondary Outcome: Seizure Frequency Per Week for All Seizure Types (Type I+II+III) Overall in the Down-titration Period
Description: Calculated as 7-day seizure frequency for all seizure types (type I+II+III). The duration of the Down-Titration Period was 3 weeks (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: During the Down-Titration Period (Week 13 to Week 15)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication. Only subjects with valid data for Type I+II+III seizure frequency per week in the down-titration period are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 27
seizures per week | 3.50 [1.75 to 13.70]

15. Secondary Outcome: Responder Rate in Partial Onset Seizures (Type I) Over the Up-titration Period
Description: A responder was defined as a subject with a >= 50% reduction in seizure frequency per week from the Baseline Period (Week 1 to Week 4) to the end of the Up-Titration Period.
Time Frame: Week 12, compared to Baseline Period (Week 1 to Week 4)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
percentage of participants | 25.8

16. Secondary Outcome: Percentage of Participants With Categorized Response to the Treatment in Partial Onset Seizures (Type I) Over the Up-titration Period
Description: Categories of percentage change in seizures from Baseline were as following: < -25%; -25% to <25%; 25% to <75%; 75% to <100%; 100%.
Time Frame: Week 12, compared to Baseline Period (Week 1 to Week 4)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
percentage of participants
  < -25% | 3.2
  -25% to < 25% | 35.5
  25% to < 75% | 51.6
  75% to <100% | 3.2
  100% | 6.5

17. Secondary Outcome: Percentage Change From Baseline in Seizure-free Days Per Week Over the Up-titration Period
Description: A day was considered seizure-free, if no seizure was reported during 24 hours.
Time Frame: Week 5 to Week 12, compared to Baseline Period (Week 1 to Week 4)
Population: The ITT set included 31 subjects, who took at least one dose of trial medication. Only subjects with valid data for seizure-free days per week over the up-titration period are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Seletracetam
Number analyzed (Participants) | 29
percentage of change | 13.80 [4.71 to 28.57]

18. Secondary Outcome: Change From Baseline in Seizure Frequency Per Week for Partial Onset Seizures (Type I) Overall in the Down-titration Period
Description: Calculated as (7-day seizure frequency during the down-titration period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)). A negative value in change from Baseline indicates a decrease in partial onset seizure frequency from Baseline. The duration of the Down-Titration Period was 3 weeks (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: During the Down-Titration Period (Week 13 to Week 15), compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 27
seizures per week | -0.96 [-3.00 to 1.41]

19. Secondary Outcome: Change From Baseline in Seizure Frequency Per Week for Partial Onset Seizures (Type I) During the Up-titration Period
Description: Calculated as (7-day seizure frequency during the up-titration period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)). A negative value in change from Baseline indicates a decrease in partial onset seizure frequency from Baseline. The duration of the Up-Titration Period was 8 weeks (Visit 3/Week 5 to Visit 7/Week 12).
Time Frame: Week 5 to Week 12, compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week | -1.14 [-4.63 to -0.50]

20. Secondary Outcome: Change From Baseline in Seizure Frequency Per Week for All Seizure Types (Types I + II + III) Overall in the Down-titration Period
Description: Calculated as (7-day seizure frequency during the down-titration period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)). A negative value in change from Baseline indicates a decrease in all seizure types frequency from Baseline. The duration of the Down-Titration Period was 3 weeks (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: Week 13 to Week 15, compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 27
seizures per week | -0.96 [-3.00 to 1.41]

21. Secondary Outcome: Change From Baseline in Seizure Frequency Per Week for All Seizure Types (Types I+II +III) Overall in the Up-titration Period
Description: Calculated as (7-day seizure frequency during the up-titration period) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)). A negative value in change from Baseline indicates a decrease in all seizure types frequency from Baseline. The duration of the Up-Titration Period was 8 weeks (Visit 3/Week 5 to Visit 7/Week 12).
Time Frame: Week 5 to Week 12, compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week | -1.14 [-4.63 to -0.50]

22. Secondary Outcome: Change From Baseline in Seizure Frequency Per Week for Partial Onset Seizures (Type I) by Visit Over the Treatment Period (Up-titration + Down-titration)
Description: Calculated as (7-day seizure frequency during the treatment period for visit n) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)). The treatment period referred to includes the period from the previous visit n-1 up to but not including the specific visit n. A negative value in change from Baseline indicates a decrease in partial onset seizure frequency from Baseline. The Overall Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: Week 5 to Week 15, compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 30
  Visit 4 (Week 5 and 6) | -1.25 [-3.00 to 0.43]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 27
  Visit 5 (Week 7 and 8) | -1.39 [-4.50 to -0.25]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 27
  Visit 6 (Week 9 and 10) | -1.25 [-5.00 to -0.45]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 30
  Visit 7 (Week 11 and 12) | -1.94 [-4.20 to -0.57]
  Visit 8 (Week 13): number analyzed (Participants) | 27
  Visit 8 (Week 13) | -1.60 [-4.75 to -0.24]
  Visit 9 (Week 14): number analyzed (Participants) | 27
  Visit 9 (Week 14) | -1.25 [-3.23 to 1.00]
  Visit 10 (Week 15): number analyzed (Participants) | 27
  Visit 10 (Week 15) | -1.50 [-3.52 to 1.62]

23. Secondary Outcome: Change From Baseline in Seizure Frequency Per Week for All Seizure Types (Types I+II+III) by Visit Over the Treatment Period (Up-titration + Down-titration)
Description: Calculated as (7-day seizure frequency during the treatment period for visit n) - (7-day seizure frequency during the Baseline Period (Week 1 to Week 4)). The treatment period referred to includes the period from the previous visit n-1 up to but not including the specific visit n. A negative value in change from Baseline indicates a decrease in all seizure types frequency from Baseline. The Overall Treatment Period consists of an 8-week Up-Titration Period (Visit 3/Week 5 to Visit 7/Week 12) and a 3-week Down-Titration Period (Visit 7/Week 13 to Visit 10/Week 15).
Time Frame: Week 5 to Week 15, compared to Baseline Period (Week 1 to Week 4)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Seletracetam
Number analyzed (Participants) | 31
seizures per week
  Visit 4 (Week 5 and 6): number analyzed (Participants) | 30
  Visit 4 (Week 5 and 6) | -1.25 [-3.00 to 0.43]
  Visit 5 (Week 7 and 8): number analyzed (Participants) | 27
  Visit 5 (Week 7 and 8) | -1.39 [-4.50 to -0.25]
  Visit 6 (Week 9 and 10): number analyzed (Participants) | 27
  Visit 6 (Week 9 and 10) | -1.25 [-5.00 to -0.45]
  Visit 7 (Week 11 and 12): number analyzed (Participants) | 30
  Visit 7 (Week 11 and 12) | -1.94 [-4.20 to -0.57]
  Visit 8 (Week 13): number analyzed (Participants) | 27
  Visit 8 (Week 13) | -1.60 [-4.75 to -0.24]
  Visit 9 (Week 14): number analyzed (Participants) | 27
  Visit 9 (Week 14) | -1.25 [-3.23 to 1]
  Visit 10 (Week 15): number analyzed (Participants) | 27
  Visit 10 (Week 15) | -1.50 [-3.52 to 1.62]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Week 1 up to Week 17
Arm/Group | Seletracetam
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 27/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seletracetam (N=31)
Sinus bradycardia (Cardiac disorders) | 1
Motion sickness (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Eye irritation (Eye disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Stomach discomfort (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Energy increased (General disorders) | 1
Fatigue (General disorders) | 2
Gait disturbance (General disorders) | 2
Irritability (General disorders) | 2
Pyrexia (General disorders) | 1
Tenderness (General disorders) | 1
Multiple allergies (Immune system disorders) | 1
Ear infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Anticonvulsant toxicity (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Tongue injury (Injury, poisoning and procedural complications) | 1
Tooth injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Platelet count decreased (Investigations) | 1
Positive Rombergism (Investigations) | 2
Red blood cell morphology abnormal (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Convulsion (Nervous system disorders) | 2
Coordination abnormal (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 4
Hypersomnia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 2
Sensory disturbance (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 10
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 1
Crying (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 1
Emotional disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Nervousness (Psychiatric disorders) | 2
Paranoia (Psychiatric disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Poor venous access (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days